CLINICAL TRIAL: NCT01673607
Title: Study of Immune Response and Liver Damage Induced by Chemotherapy for Liver Metastases of Colorectal Cancer
Acronym: METAHEP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: METAHEP
Record Dates: First submitted 2012-02-13; First posted 2012-08-28 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Resectable Hepatic Metastases of Colorectal Cancer

INTERVENTIONS:
Procedure: Biopsie liver

SUMMARY:
The immune response at primary tumor has a major role in the prognosis of colorectal cancer (CRC). Some studies suggest a prognosis value of cytotoxic T cell and memory T cells at primary tumor greater than tumoral stage. There is no work in the literature that has examined the prognosis value of the immune response in liver metastases. To study immune cells (histology) and inflammatory response (cytokines) in liver metastases is a challenge to understand the effectiveness of chemotherapy used in this situation.

The chemotherapy used in liver metastases of colorectal cancer also have effects on non-tumoral liver tumor and therefore can interfere with postoperative complications of hepatic resection. Sinusoidal dilatation is present in 20% to 80% of patients who received oxaliplatin before hepatectomy. Steatosis is frequently observed after administration of 5-FU alone or in combination with irinotecan. This steatosis may also be accompanied by inflammatory lesions (steatohepatitis), especially after administration of oxaliplatin or irinotecan and is associated with increased postoperative mortality. The hepatic toxicity of new biological agents is not well known (cetuximab and bevacizumab). The mechanisms of chemotherapy-induced toxicities are currently unknown. The main objective is to analyze the profile of the immune response in liver metastases of CRC and find the link with the radiological response. Measurements will be made by quantitative RT-PCR on frozen liver biopsies. Secondary objective is to seek a correlation between the histological lesions induced by chemotherapy and non-invasive tests for liver fibrosis. The secondary endpoints are rate of immune cells, histologic response (percentage of tumor necrosis), disease-free survival, the non-invasive test of fibrosis, the chemotherapy-induced liver injury, cytokines and circulating angiogenic factors.

ELIGIBILITY:
Inclusion Criteria:

Patient older than 18 years.

* Patients with histologically proven colorectal cancer with resectable or potentially resectable liver metastases.
* First line chemotherapy alone or combination with intravenous 5FU, oral 5FU (capecitabine), oxaliplatin, irinotecan, cetuximab, panitumumab or bevacizumab (LV5FU2, XELODA, FOLFIRI, FOLFOX, XELOX, XELIRI alone or in combination with either cetuximab or panitumumab or bevacizumab).
* Signature of informed consent.
* Patient affiliated to French Social Security.

Exclusion Criteria:

Patients taking immunosuppressive therapy.

* Lack of measurable tumoral target.
* Patients with a contre-indication of all chemotherapy used: oxaliplatin, irinotecan, fluorouracil, capecitabine, cetuximab, panitumumab, bevacizumab.
* Patients hospitalized without consent.
* Patients in emergency situations.
* Patients under guardianship.
* Patients deprived of their liberty by judicial or administrative procedure.
* Pregnant or nursing women, women without effective contraception.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, France